CLINICAL TRIAL: NCT06463873
Title: A Pilot Study of OmniGraft in Simultaneous Pancreas Kidney Recipients
Brief Title: Study of OmniGraft in Simultaneous Pancreas Kidney Recipients
Status: Terminated | Type: Observational
Why Stopped: The sponsor suspended the financial support.
Sponsor: University of Miami (Other)
Collaborators: Eurofins Lancaster Laboratories (Unknown)
Responsible Party: Principal Investigator, Mariella Ortigosa Goggins, Associate Professor of Clinical, University of Miami
Other Study IDs: 20221147
Record Dates: First submitted 2024-06-10; First posted 2024-06-18 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-10

CONDITIONS: Kidney Transplant; Complications; Pancreas Disease
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Omnigraft 3 month - 1 year Group 1: Subjects will be enrolled between 2 months and 1 year post Simultaneous Pancreas Kidney (SPK) transplant. Blood sample to test Omnigraft will be collected monthly month or every 3 months depending on the enrollment time, time of rejection, or when a biopsy is done.
- Omnigraft 1 year - 3 years Group 2: Subjects will be enrolled between 12 months and 3 year post SPK transplant. Blood sample to test Omnigraft will be collected every 3 months, at the time of rejection or when a biopsy is done.
- Omnigraft 10 years Group 3: Subjects will be enrolled between 3 years to 10 years post SPK transplant. Then, blood samples to test Omnigraft will be collected every 3 months, time of rejection or when a biopsy is done.

SUMMARY:
The purpose of this research is learn about how OmniGraf works in kidney pancreas transplant patients. Also, to analyze the performance characteristics of OmniGrafTM (TruGraf Gene Expression Profiling (GEP) and T Cell Receptor Alpha Constant (TRAC) dd-cfDNA) in a population of simultaneous kidney pancreas transplants as a part of routine surveillance, as well as a part of the workup for patients clinically suspected to have rejection of the kidney and/or pancreas.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult (≥18 years old) with a history of simultaneous pancreas kidney transplant between 3 months and 1 year prior to enrollment (cohort 1) or at the time of presentation for "for-cause" biopsy
2. Adults able to consent
3. Bladder or enteric drained
4. Type 1 or Type 2 DM

Exclusion Criteria:

1. Recipient of an organ transplant other than a simultaneous pancreas kidney transplant
2. Known to be pregnant
3. Known to be infected with Human Immunodeficiency Virus with actively replicating HIV virus
4. Active BK viremia with >100,000 copies or biopsy proven BK nephropathy
5. Participation in other biomarker studies
6. Pancreas transplant alone
7. Re-transplantation, unless both organs have been removed prior to or at the time of the retransplant procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Simultaneous kidney pancreas transplant who are treated at the Miami Transplant Institute
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Number of participants that underwent SPK transplant | Up to 3 years
  Number of participants that underwent SPK transplant measured by Omnigraft testing. The Omnigraft test includes TruGraf GEP and TRAC dd-cfDNA.

CONTACTS AND LOCATIONS:
Overall Officials: Mariella Ortigosa-Goggins, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Miami Transplant Institute 1801 NW 9th Ave, Miami, Florida
  - University of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No